CLINICAL TRIAL: NCT01003210
Title: Homeopathic Ear Drops for Children With Otitis Media Study
Brief Title: Homeopathic Ear Drops for Otitis Media Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, James Taylor, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 37011
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Otitis Media
Keywords: otitis media; children; homeopathy
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homeopathic ear drops (Experimental): Commercially available homeopathic ear drops
  Interventions: Drug: Hyland's earache drops
- standard therapy (No Intervention): standard therapy for otitis media, no ear drops

INTERVENTIONS:
Drug: Hyland's earache drops — 3-4 drops in affected ear 3 times a day as needed for up to 5 days
  Arms: Homeopathic ear drops

SUMMARY:
The purpose of this study is to determine if a commercially available homeopathic ear drop preparation is effective in reducing symptoms in children 6 months - 11 years old with acute otitis media in whom the health care provider has recommended that antibiotics not be immediately administered. A total of 150 study patients with otitis media will be randomized to receive homeopathic ear drops, or no ear drops, in addition to receiving standard care. It is postulated that children using the ear drops will have more rapid resolution of symptoms and need fewer antibiotics than those randomized to not receive the ear drops.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 11 years old
* Diagnosed with otitis media by clinician at participating clinic
* Clinician determines that a "watch and wait" antibiotic prescription treatment plan is optimal management

Exclusion Criteria:

* Antibiotic treatment during past 7 days
* Homeopathic treatment within past 30 days
* History of serious chronic illness (e.g. diabetes, autoimmune disease, cystic fibrosis
* Perforated tympanic membrane
* Immediate antibiotic treatment plan decided by examining clinician

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Mercer Island Pediatric Associates, Mercer Island, Washington
  - Valley Children's Clinic, Renton, Washington
  - University of Washington Medical Center-Roosevelt Pediatric Care Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homeopathic Ear Drops | Standard Therapy
Started | 105 | 105
Completed | 104 | 102
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Children 6 months - 11 years old diagnosed with acute otitis media and managed with a delayed antibiotic treatment approach
Groups:
- Total: Total of all reporting groups
Arm/Group | Homeopathic Ear Drops | Standard Therapy | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 105 | 105 | 210
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.9 (2.8) | 4.2 (2.6) | 4.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 77 | 128
  Male | 54 | 28 | 82
Region of Enrollment [Number; unit: participants]
  United States | 105 | 105 | 210

OUTCOME MEASURES:

1. Primary Outcome: Severity of Symptoms of Otitis Media
Description: Ear Treatment Group - 5 scores. Parent rated severity of otitis media symptoms including fever, earache, irritability, feeding and sleeping. Each symptom rated 0, 4 or 7. Total scores range 0 (least symptoms) to 35 most symptom. ETG-5 scores collected 12-15 days after enrollment
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Homeopathic Ear Drops | Standard Therapy
Number analyzed (Participants) | 101 | 99
units on a scale | 2.0 (4.5) | 2.0 (3.8)

2. Primary Outcome: Administration of Antibiotics
Description: Number of participants who filled antibiotic prescription (or called back for promised antibiotic prescription) after being diagnosed with acute otitis media at index visit.
Time Frame: 15 days
Measure: Number; unit: participants
Arm/Group | Homeopathic Ear Drops | Standard Therapy
Number analyzed (Participants) | 104 | 102
participants | 28 | 42

3. Secondary Outcome: Side Effects From Study Remedy
Description: Any "other symptoms" reported by parents in logbooks. Logbooks were returned by 72/105 participants randomized to the homeopathic ear drops group and 78 of those randomized to standard therapy alone.
Time Frame: 15 days
Population: The number of participants analyzed includes only those whose parents returned logbooks.
Measure: Number; unit: participants
Arm/Group | Homeopathic Ear Drops | Standard Therapy
Number analyzed (Participants) | 72 | 78
participants
  vomit | 4 | 5
  rash | 3 | 11
  diarrhea | 5 | 6
  "hyper" behavior | 6 | 10
  headache | 9 | 10
  lethargy | 15 | 23
  other symptom reported | 14 | 23
  decreased hearing | 1 | 0
  "plugged" ears | 1 | 0
  redness around ear with drops | 1 | 0
  ear popping | 1 | 0

ADVERSE EVENTS:
Description: Adverse data were not collected on 4 children including 1 randomized to the ear drop group and 3 receiving standard therapy alone.
Arm/Group | Homeopathic Ear Drops | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/102
Other Adverse Events (participants affected / at risk) | 58/104 | 88/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Homeopathic Ear Drops (N=104) | Standard Therapy (N=102)
vomit (Gastrointestinal disorders) | 4 (5) | 5 (8)
rash (Skin and subcutaneous tissue disorders) | 3 (8) | 11 (22)
diarrhea (Gastrointestinal disorders) | 5 (14) | 6 (15)
"hyper" behavior (Psychiatric disorders) | 9 (22) | 10 (16)
Headache (General disorders) | 9 (22) | 10 (16)
lethargy (General disorders) | 15 (27) | 23 (58)
Others (General disorders) | 14 (48) | 23 (83)
decreased hearing (Ear and labyrinth disorders) | 1 (4) | 0 (0)
ear plugging (Ear and labyrinth disorders) | 1 (2) | 0 (0)
ears popping (Ear and labyrinth disorders) | 1 (1) | 0 (0)
redness around ear (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Initially planned sample size --150. Study size was increased after analysis of initial data found a non-significant trend between antibiotic fill rates in the homeopathic ear drop and standard therapy treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No